CLINICAL TRIAL: NCT03485638
Title: Assessment and Prediction of Cetuximab-Induced Hypersensitivity Reactions Using Cetuximab Specific IgE Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0811
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Tumor Disease Including Colorectal Cancer; Head & Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cetuximab administration

SUMMARY:
1. Background Cetuximab (trade name Erbitux) is a murine-human chimeric monoclonal antibody to human epidermal growth factor receptor (EGFR). This drug has been used as a treatment for colorectal cancer and head and neck cancer. It is known that allergic reactions can occur in more than 5% of the patients, although the side effects are relatively low compared with other chemotherapeutic agents. It is known that cetuximab can induce hypersensitivity even at the first administration, unlike other anticancer drugs. In this study, we aimed to establish a model to predict patients with hypersensitivity reaction before administration of cetuximab and to provide safe chemotherapy.
2. Recruitment method and consent procedure The study is designed for analysis patients scheduled for administration of cetuximab for the first time. Patients matching the selection and exclusion criteria with voluntary agreement to the study will be enrolled. Enrolled patients will be tested for skin prick test and serum sIgE before cetuximab administration.

DETAILED DESCRIPTION:
* Acquisition of agreement Agreement, explanation, and consent form for study of human derived sample those that approved by the IRB are obtained from patients who prospectively voluntarily participate in the study and provide human derived sample.
* Observation and evaluation values

  ① Serum Cetuximab-specific IgE measurement (ImmunoCAP, conventional ELISA) before administration of cetuximab

  ② Cetuximab Skin test using before cetuximab administration

  ③ Clinical symptoms after cetuximab administration through chart review (vital signs, occurrence of adverse drug reaction)

  ④ Check patient's underlying disease and allergy history
* Statistical analysis method Chi-square test, Fisher's exact test, Student t-test, Mann-Whitney test, Logistic regression test, Cox's regression test, and ROC curve will be used

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 18 years of age
* Patients scheduled for cetuximab administration according to standard treatment guidelines for the treatment of underlying tumor disease.

Exclusion Criteria:

* Patients who did not consent to the study voluntarily after IRB approval
* Persons who are vulnerable (including persons with disabilities, lack of physician capacity, pregnant status, persons who are accommodated in facilities, etc.)
* Those who can not read and understand the agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for Cetuximab administration according to standard treatment guidelines for the treatment of underlying tumor disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-11-04 (Actual); Primary Completion 2020-11-03 (Estimated); Study Completion 2020-11-03 (Estimated)

PRIMARY OUTCOMES:
Hypersensitivity reaction after cetuximab administration | Within 4 weeks after first administration
  Adverse drug reaction after Cetuximab administration includes severe systemic allergic reaction such as anaphylaxis, urticaria, skin rash, dyspnea, shock and mental change.

SECONDARY OUTCOMES:
Cetuximab specific IgE | within 4 weeks after first administration
  Cetuximab specific IgE measured by ImmunoCAP assay, ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Allergy and Immunology, Department of Internal Medicine, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George TJ Jr, Laplant KD, Walden EO, Davis AB, Riggs CE, Close JL, George SN, Lynch JW. Managing cetuximab hypersensitivity-infusion reactions: incidence, risk factors, prevention, and retreatment. J Support Oncol. 2010 Mar-Apr;8(2):72-7. PMID 20464886
- [Background] Hansen NL, Chandiramani DV, Morse MA, Wei D, Hedrick NE, Hansen RA. Incidence and predictors of cetuximab hypersensitivity reactions in a North Carolina academic medical center. J Oncol Pharm Pract. 2011 Jun;17(2):125-30. doi: 10.1177/1078155209360853. Epub 2010 Feb 10. PMID 20147576
- [Background] Chung CH, Mirakhur B, Chan E, Le QT, Berlin J, Morse M, Murphy BA, Satinover SM, Hosen J, Mauro D, Slebos RJ, Zhou Q, Gold D, Hatley T, Hicklin DJ, Platts-Mills TA. Cetuximab-induced anaphylaxis and IgE specific for galactose-alpha-1,3-galactose. N Engl J Med. 2008 Mar 13;358(11):1109-17. doi: 10.1056/NEJMoa074943. PMID 18337601
- [Background] Pointreau Y, Commins SP, Calais G, Watier H, Platts-Mills TA. Fatal infusion reactions to cetuximab: role of immunoglobulin e-mediated anaphylaxis. J Clin Oncol. 2012 Jan 20;30(3):334; author reply 335. doi: 10.1200/JCO.2011.38.4701. Epub 2011 Dec 12. No abstract available. PMID 22162592
- [Background] Mariotte D, Dupont B, Gervais R, Galais MP, Laroche D, Tranchant A, Comby E, Bouhier-Leporrier K, Reimund JM, Le Mauff B. Anti-cetuximab IgE ELISA for identification of patients at a high risk of cetuximab-induced anaphylaxis. MAbs. 2011 Jul-Aug;3(4):396-401. doi: 10.4161/mabs.3.4.16293. Epub 2011 Jul 1. PMID 21654207
- [Background] Maier S, Chung CH, Morse M, Platts-Mills T, Townes L, Mukhopadhyay P, Bhagavatheeswaran P, Racenberg J, Trifan OC. A retrospective analysis of cross-reacting cetuximab IgE antibody and its association with severe infusion reactions. Cancer Med. 2015 Jan;4(1):36-42. doi: 10.1002/cam4.333. Epub 2014 Oct 9. PMID 25296628
- [Background] Jerath MR, Kwan M, Kannarkat M, Mirakhur B, Carey L, Valgus J, Platts-Mills TA, Tarrant TK. A desensitization protocol for the mAb cetuximab. J Allergy Clin Immunol. 2009 Jan;123(1):260-2. doi: 10.1016/j.jaci.2008.09.046. Epub 2008 Nov 20. No abstract available. PMID 19022494